CLINICAL TRIAL: NCT00407732
Title: Overcoming Neuropsychiatric Barriers to the Treatment of Hepatitis C
Brief Title: Overcoming Psychiatric Barriers to the Treatment of Hepatitis C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Donna Evon, Assistant Professor of Medicine, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 05-2944 PEG228
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Hepatitis C; Substance Use Disorders; Mental Disorder
Keywords: hepatitis C; mental disorder; substance use; psychosocial intervention
MeSH Terms: conditions — Hepatitis C; Substance-Related Disorders; Mental Disorders | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SC (No Intervention): standard care
- INT (Experimental): psychosocial intervention
  Interventions: Behavioral: psychosocial intervention

INTERVENTIONS:
Behavioral: psychosocial intervention — motivational enhancing case management intervention
  Arms: INT

SUMMARY:
The purpose of this study is to develop and evaluate a 9-month psychosocial intervention that will assist patients with hepatitis C in overcoming barriers that prevent them from becoming appropriate candidates for interferon therapy.

DETAILED DESCRIPTION:
The purpose of this study is to develop and evaluate a 9-month psychosocial intervention that will assist patients with hepatitis C in overcoming barriers that prevent them from becoming appropriate candidates for interferon therapy. Patients who have been deferred from therapy due to mental health or substance abuse issues will work with the team psychologist on following through with the hepatologist's treatment recommendations that would lead to becoming eligible for interferon therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient has confirmed diagnosis of HCV;
* Patient has expressed an interest in undergoing interferon treatment;
* Patient is deferred from interferon therapy for psychiatric, alcohol use, or other psychosocial issues;
* Patient must be completely medically cleared by the hepatologist with no outstanding medical conditions that would deem them ineligible from treatment;
* Patient must have only psychiatric issues and/or substance use issues; but otherwise no other contraindications for treatment.

Exclusion Criteria:

* Patient has a diagnosis of schizophrenia, psychosis;
* Patient resides in a psychiatric residential facility;
* Patient attempted suicide in the past five years;
* Patient is a current intravenous drug user;
* Patient is cognitively or decisionally-impaired due to brain disease or injury;
* Patient has advanced liver disease that precludes them from interferon treatment;
* Patient has other medical comorbidities that may exclude them from interferon treatment;
* Patient does not want to pursue interferon treatment at the present time;
* Patient has significant financial constraints, such as no insurance or homelessness, that would prevent them acquiring mental health or substance abuse services;
* No access to telephone service;
* Non-English speaking.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-01; Primary Completion 2010-02 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Whether or not the patient is deemed an appropriate candidate for interferon therapy at the end of the 9-month intervention. | 3-, 6-, and 9-months

CONTACTS AND LOCATIONS:
Overall Officials: Donna M Evon, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Unversity of North Carolina, Chapel Hill, North Carolina, United States